CLINICAL TRIAL: NCT01518153
Title: Phase 2 Study of Planned Donor Lymphocyte Infusion After Reduced Intensity Allogeneic Stem Cell Transplantation
Brief Title: Planned Donor Lymphocyte Infusion (DLI) After Allogeneic Stem Cell Transplantation (SCT)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Objectives not met.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-1104; NCI-2012-00131 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-01-23; First posted 2012-01-25 (Estimated); Results first posted 2016-03-17 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-02

CONDITIONS: Leukemia; Lymphoma; Myeloma; Myeloproliferative Diseases
Keywords: Blood and Marrow Transplantation; Lymphoma; Myeloma; Myeloproliferative Diseases; Leukemia; Myelodysplastic syndrome; MDS; Hodgkin disease; Multiple myeloma; Fludarabine; Fludarabine Phosphate; Fludara; Melphalan; Alkeran; Tacrolimus; Prograf; Methotrexate; G-CSF; Filgrastim; NeupogenTM; Donor Lymphocyte Infusion; DLI; Allogeneic Stem Cell Transplantation; Graft-vs-host disease; GvHD; T-lymphocytes; T-cells; Alemtuzumab; CAMPATH-1H; Campath
MeSH Terms: conditions — Leukemia; Lymphoma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Hodgkin Disease; Multiple Myeloma; Graft vs Host Disease | interventions — fludarabine; fludarabine phosphate; Melphalan; Alemtuzumab; Tacrolimus; Methotrexate; Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Dose Donor T-Cells (Experimental): Fludarabine 40 mg/m^2 by vein on Day -6 to -3. Melphalan 140 mg/m^2 by vein on Day -2. Alemtuzumab 50 mg by vein on Day -1. Reduced intensity stem cell transplant on Day 0. Planned Donor Lymphocyte Infusion CD3+ cells: 3 * 106 CD3+ cells/kg between Day +56 and +64. Tacrolimus 0.015 mg/kg by vein as a 24 hour continuous infusion daily adjusted to achieve a therapeutic level of 5-15 ng/ml (target is 10 ng/ml). Tacrolimus is changed to oral dosing when tolerated. Tapering should start on approximately Day +24 with intention to be completely off drug by approximately Day +35. Methotrexate 5 mg/m2 dosed based on actual body surface area and administered intravenously on days +1, +3, +6. G-CSF 5 mcg/kg/day subcutaneously beginning on Day +7, and continuing until absolute neutrophil count (ANC) is > 500 * 10/L for 3 consecutive days.
  Interventions: Drug: Fludarabine; Drug: Melphalan; Drug: Alemtuzumab; Procedure: Stem Cell Infusion; Drug: Tacrolimus; Drug: Methotrexate; Drug: G-CSF; Procedure: Low Dose Donor T-Cells
- High Dose Donor T-Cells (Experimental): Fludarabine 40 mg/m^2 by vein on Day -6 to -3. Melphalan 140 mg/m^2 by vein on Day -2. Alemtuzumab 50 mg by vein on Day -1. Reduced intensity stem cell transplant on Day 0. High Dose Donor T-Cells Planned Donor Lymphocyte Infusion CD3+ cells: 1 * 107 CD3+ cells/kg between Day +56 and +64. Tacrolimus 0.015 mg/kg by vein as a 24 hour continuous infusion daily adjusted to achieve a therapeutic level of 5-15 ng/ml (target is 10 ng/ml). Tacrolimus is changed to oral dosing when tolerated. Tapering should start on approximately Day +24 with intention to be completely off drug by approximately Day +35. Methotrexate 5 mg/m2 dosed based on actual body surface area and administered intravenously on days +1, +3, +6. G-CSF 5 mcg/kg/day subcutaneously beginning on Day +7, and continuing until absolute neutrophil count (ANC) is > 500 * 10/L for 3 consecutive days.
  Interventions: Drug: Fludarabine; Drug: Melphalan; Drug: Alemtuzumab; Procedure: Stem Cell Infusion; Drug: Tacrolimus; Drug: Methotrexate; Drug: G-CSF; Procedure: High Dose Donor T-Cells

INTERVENTIONS:
Drug: Fludarabine — 40 mg/m^2 by vein on Day -6 to -3.
  Other Names: Fludarabine Phosphate; Fludara
Drug: Melphalan — 140 mg/m^2 by vein on Day -2.
  Other Names: Alkeran
Drug: Alemtuzumab — 50 mg by vein on Day -1.
  Other Names: CAMPATH-1H; Campath
Procedure: Stem Cell Infusion — Reduced intensity stem cell transplant on Day 0.
Drug: Tacrolimus — 0.015 mg/kg by vein as a 24 hour continuous infusion daily adjusted to achieve a therapeutic level of 5-15 ng/ml (target is 10 ng/ml). Tacrolimus is changed to oral dosing when tolerated. Tapering should start on approximately Day +24 with intention to be completely off drug by approximately Day +35.
  Other Names: Prograf
Drug: Methotrexate — 5 mg/m2 dosed based on actual body surface area and administered intravenously on days +1, +3, +6.
Drug: G-CSF — 5 mcg/kg/day subcutaneously beginning on Day +7, and continuing until absolute neutrophil count (ANC) is > 500 * 10/L for 3 consecutive days.
  Other Names: Filgrastim; NeupogenTM
Procedure: Low Dose Donor T-Cells — Planned Donor Lymphocyte Infusion CD3+ cells: 3 * 106 CD3+ cells/kg between Day +56 and +64.
  Arms: Low Dose Donor T-Cells
Procedure: High Dose Donor T-Cells — Planned Donor Lymphocyte Infusion CD3+ cells: 1 * 107 CD3+ cells/kg between Day +56 and +64.
  Arms: High Dose Donor T-Cells

SUMMARY:
The goal of this clinical research study is to learn what dose of a kind of immune cell called T-lymphocytes (T-cells) given as a donor infusion about 8-9 weeks after a stem cell transplant has the best results. The safety of this treatment will also be studied. This will be tested in patients with leukemia, MDS, lymphoma, Hodgkin disease, and multiple myeloma. These results are measured as helping to control the disease without severe graft-versus-host disease (GvHD). GvHD is when transplanted donor tissue attacks the tissues of the recipient's body.

Fludarabine, melphalan, and alemtuzumab are commonly given before stem cell transplants:

* Fludarabine is designed to interfere with the DNA (genetic material) of cancer cells, which may cause the cancer cells to die.
* Melphalan is designed to bind to the DNA of cells, which may cause cancer cells to die.
* Alemtuzumab is designed to weaken the immune system and reduce the risk of rejection of the transplant and graft-vs-host disease (GvHD).

The donor infusion of T-cells is designed to help restore the immune system after the transplant, cause an immune reaction against the cancer, and reduce the risk of the cancer coming back.

DETAILED DESCRIPTION:
Study Groups:

If you agree to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups involving the dose of T-cells in the donor lymphocyte infusion.

* Group 1 will receive a low dose of donor T-cells.
* Group 2 will receive a higher dose of donor T-cells than Group 1.

Both you and your study doctor will know which group you are in. Both groups will have a stem cell transplant. The stem cells will be given by vein. The cells will travel to your bone marrow where they are designed to make healthy, new blood cells after several weeks.

Study Drug Administration:

Patients receive fludarabine, melphalan and alemtuzumab to kill malignant cells and suppress immunity to prevent rejection of the stem cell transplant. The day you receive the stem cells is called Day 0. The days before you receive your stem cells are called minus days. The days after you receive the stem cells are called plus days.

On Day -7, you will be admitted to the hospital and given fluids by vein to hydrate you.

On Days -6 through -3, you will receive fludarabine by vein over 1 hour each day.

On Day -2, you will receive melphalan by vein over 30 minutes.

On Day -1, you will receive alemtuzumab by vein over 2 hours.

On Day 0, you will receive the stem cell transplant as a cell infusion by vein.

After the transplant, you will receive tacrolimus and methotrexate. At first, you will receive tacrolimus as a continuous (nonstop) infusion until you are able to take it by mouth. You will then take tacrolimus by mouth 2 times a day for about 5 weeks and then your doctor will tell you how to taper it off (gradually stop taking it). On Days 1, 3, and 6 after the transplant, you will receive methotrexate by vein over 30 minutes.

You will receive filgrastim as an injection under the skin 1 time a day, starting 1 week after the transplant, until your blood cell levels return to normal. Filgrastim is designed to help with the growth of white blood cells.

Between Day +56 and +64, if you are in stable medical condition and have not developed GvHD, you will receive a donor lymphocyte infusion containing T-cells by vein over 10-30 minutes. You will receive Benadryl (diphenhydramine) by vein over 15 minutes before the infusion to lower the risk of an allergic reaction.

Study Visits:

Before the T-cell infusion:

* You will have a physical exam, including measurement of your vital signs (blood pressure, heart rate, temperature, and breathing rate).
* You will be asked about how you are feeling and about any side effects you may be having.
* Blood (about 2 teaspoons) will be drawn to see how well the transplant has "taken".
* You will have a bone marrow aspiration and biopsy to check the status of the disease, if your doctor thinks it is needed. To collect a bone marrow aspiration/biopsy, an area of the hip or other site is numbed with anesthetic, and a small amount of bone marrow and bone is withdrawn through a large needle.

After the T-cell infusion, you will have a physical exam every week for at least 6 weeks.

About 3, 6, and 12 months after the transplant:

* You will have a physical exam, including measurement of your vital signs.
* You will be asked about how you are feeling and about any side effects you may be having.
* Blood (about 4 tablespoons) will be drawn for routine tests and to check the level of the infused T-cells, for immune function tests, and to check the status of the disease.
* You will have a bone marrow aspiration, blood tests and CT scans as medically necessary to check the status of the disease, if your doctor thinks it is needed.

During the study, you will have blood draws (about 2 teaspoons) and urine will be collected for routine tests, to check your blood counts, kidney and liver function, and/or to check for infections as often as the doctor thinks is needed during this time.

Length of Treatment:

You will be off study after your 12-month follow-up visit. You will be taken off study early if you have graft failure (the donor cells did not "take") or if the cancer comes back and needs another treatment.

This is an investigational study. Melphalan, fludarabine, and alemtuzumab are FDA approved and commercially available for the treatment of blood cancers. Donor T-cell infusions are commonly used to treat blood cancers that come back after a stem cell transplant. The investigational part of this study is to find the best dose of T-cells that are given with the goal of helping to prevent the cancer from coming back.

Up to 56 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/= 18 years and </= 65 years with one of the following: a. Acute leukemia past first remission, in first or subsequent relapse, in second or greater remission. Patients in first remission should have intermediate or high cytogenetic risk factors or flt3 mutation. Patients with primary induction failure or relapse are eligible if they have <10% bone marrow blasts, and no circulating blasts. b. Myelodysplastic syndrome with intermediate or high risk IPSS score, or treatment related MDS. c. CML resistant to tyrosine kinase inhibitor treatment in a first or subsequent chronic phase, or in accelerated phase. d. CLL, Lymphoma or Hodgkin's disease which has failed to achieve remission or recurred following initial chemotherapy. Patients must have at least a PR to salvage therapy, or low bulk untreated relapse (<2 cm largest mass). e. Multiple myeloma which has relapsed or progressed and has achieved a partial response to salvage chemotherapy.
2. Patients must have one of the following donor types identified and willing to donate: a. Related donor, HLA-matched for HLA-A, -B, C and DR matched or, b. Matched Unrelated Donor (MUD), HLA-matched for HLA A, B, C and DRB1 using allele level typing.
3. Performance score of at least 80% by Karnofsky or performance score 0 to 2 (ECOG).
4. Estimated creatinine clearance >40 ml/min (based on serum creatinine)
5. Bilirubin <1.5 mg/dl except for Gilbert's disease.
6. ALT < 300 IU/ml d.
7. Left ventricular ejection fraction equal or greater than 40%.
8. Pulmonary function test (PFT) demonstrating a diffusion capacity (corrected for hemoglobin) of least 50% predicted.
9. Patient or patient's legal representative able to sign informed consent.

Exclusion Criteria:

1. Patients who have had prior autologous transplants or prior allogeneic transplants are not eligible.
2. Uncontrolled active infection.
3. Positive Beta HCG test in a woman with child bearing potential, defined as not post-menopausal for 12 months or no previous surgical sterilization.
4. Women of child bearing potential not willing to use an effective contraceptive measure while on study.
5. Subject has known sensitivity to any of the products that will be administered during the study.
6. Patients who are HIV seropositive.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard E. Champlin, MD,BS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: February 6, 2012 to February 27, 2014. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Sixteen participants have been treated on study and were evaluable for treatment response. Out of 16, 7 participants met the criteria to receive planned Donor Lymphocyte Infusion (DLI). 9 participants did not meet the criteria to receive randomized planned DLI.
Groups:
- Stem Cell Infusion: Fludarabine 40 mg/m^2 intravenous (IV) administered from Day -6 to -3, Melphalan 140 mg/m^2 IV on Day -2 and Alemtuzumab 50 mg IV on Day -1. Day 0 Stem Cell infusion: Fresh or cryopreserved peripheral blood progenitor cells infused.
- Low Dose Donor T-Cells: Fludarabine 40 mg/m^2 intravenous (IV) administered from Day -6 to -3, Melphalan 140 mg/m^2 IV on Day -2 and Alemtuzumab 50 mg IV on Day -1. Day 0 Stem Cell infusion: Fresh or cryopreserved peripheral blood progenitor cells infused. Planned Donor Lymphocyte Infusion CD3+ cells: 1*10^6 CD3+ cells/kg between Day +56 & +64. Tacrolimus 0.015 mg/kg IV as continuous infusion daily to achieve therapeutic level of 5-15 ng/ml (target 10 ng/ml). Tacrolimus changed to oral dosing, tapering approximately Day +35 to off by Day +42. Methotrexate 5 mg/m^2 administered IV days +1, +3, +6. G-CSF 5 mcg/kg/day subcutaneously beginning Day +7, continuing until absolute neutrophil count (ANC)> 500*10/L for 3 consecutive days.
- High Dose Donor T-Cells: Fludarabine 40 mg/m^2 intravenous (IV) administered from Day -6 to -3, Melphalan 140 mg/m^2 IV on Day -2 and Alemtuzumab 50 mg IV on Day -1. Day 0 Stem Cell infusion: Fresh or cryopreserved peripheral blood progenitor cells infused. Planned Donor Lymphocyte Infusion CD3+ cells: 3*10^6 CD3+ cells/kg between Day +56 & +64. Tacrolimus 0.015 mg/kg IV as continuous infusion daily to achieve therapeutic level of 5-15 ng/ml (target 10 ng/ml). Tacrolimus changed to oral dosing, tapering approximately Day +35 to off by Day +42. Methotrexate 5 mg/m^2 administered IV days +1, +3, +6. G-CSF 5 mcg/kg/day subcutaneously beginning Day +7, continuing until absolute neutrophil count (ANC)> 500*10/L for 3 consecutive days.
Period: Stem Cell Transplant
Arm/Group | Stem Cell Infusion | Low Dose Donor T-Cells | High Dose Donor T-Cells
Started | 16 | 0 | 0
Completed | 7 | 0 | 0
Not Completed | 9 | 0 | 0
Not completed — Active graft-vs-host disease (GvHD) | 5 | 0 | 0
Not completed — Death | 2 | 0 | 0
Not completed — Secondary graft failure | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Period: Donor Lymphocyte Infusion
Arm/Group | Stem Cell Infusion | Low Dose Donor T-Cells | High Dose Donor T-Cells
Started | 0 | 3 | 4
Completed | 0 | 1 | 3
Not Completed | 0 | 2 | 1
Not completed — Death | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Stem Cell Transplant + Donor Lymphocyte Infusion: Fludarabine 40 mg/m^2 intravenous (IV) administered from Day -6 to -3, Melphalan 140 mg/m^2 IV on Day -2 and Alemtuzumab 50 mg IV on Day -1. Day 0 Stem Cell infusion: Fresh or cryopreserved peripheral blood progenitor cells infused. Planned Donor Lymphocyte Infusion CD3+ cells: 1 x 10^6 CD3+ cells/kg or 3 x 10^6 CD3+ cells/kg between Day +56 & +64. Tacrolimus 0.015 mg/kg IV as continuous infusion daily to achieve therapeutic level of 5-15 ng/ml (target 10 ng/ml). Tacrolimus changed to oral dosing, tapering approximately Day +35 to off by Day +42. Methotrexate 5 mg/m^2 administered IV days +1, +3, +6. G-CSF 5 mcg/kg/day subcutaneously beginning Day +7, continuing until absolute neutrophil count (ANC)> 500*10/L for 3 consecutive days.
Arm/Group | Stem Cell Transplant + Donor Lymphocyte Infusion
Number analyzed (Participants) | 16
Age, Continuous [Median (Full Range); unit: years] | 58 [35 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Success Rate
Description: Success rate defined as alive, engrafted without grade 3 or 4 GvHD or relapse at day 100 post allogeneic stem cell transplantation followed by donor lymphocyte infusion (DLI).
Time Frame: 100 days
Population: Sixteen participants have been treated on study and were evaluable for treatment response. Out of 16, 7 participants met the criteria to receive planned DLI. 9 participants did not meet the criteria to receive randomized planned DLI.
Measure: Number; unit: participants
Arm/Group | Low Dose Donor T-Cells | High Dose Donor T-Cells
Number analyzed (Participants) | 3 | 4
participants | 1 | 3

2. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival is defined as the interval between day of transplant and day of death.
Time Frame: Every 3 months until day of death
Population: Sixteen participants have been treated on study and were evaluable for treatment response. Out of 16, 7 participants met the criteria to receive planned DLI.
Measure: Median (Full Range); unit: days
Arm/Group | Stem Cell Transplant + Donor Lymphocyte Infusion
Number analyzed (Participants) | 16
days | 246 [26 to 504]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the start of preparative regimen up to discontinuation of study treatment. Overall collection period: March 30, 2012 to April 15, 2014.
Arm/Group | Stem Cell Infusion | Low Dose Donor T-Cells | High Dose Donor T-Cells
Serious Adverse Events (participants affected / at risk) | 9/9 | 2/3 | 4/4
Other Adverse Events (participants affected / at risk) | 9/9 | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stem Cell Infusion (N=9) | Low Dose Donor T-Cells (N=3) | High Dose Donor T-Cells (N=4)
Death (General disorders) | 5 (5) | 2 (2) | 1 (1)
Idiopathic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Secondary Graft Failure (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Enterococcus Faecium Stool Infection (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Parvovirus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Disseminated Cytomegalovirus Infections (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pseudomonas Bacteremia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral Exanthem (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) — Suspected due to preparatory regimen
Liver GvHD (Hepatobiliary disorders) | 0 (0) | 1 (1) | 3 (4)
Pneumocystis Jiroveci (PCP) Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fusarium Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Nocardiosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pseudomonas Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenic Fevers (General disorders) | 1 (1) | 0 (0) | 1 (1)
Staphylococcus Epidermidis Bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Candida Albicans (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Escherichia Coli Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Staphylococcus Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Acute Tubular Necrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) — Pre-existing renal insufficiency
Pseudomonas Tracheitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Anoxic Brain Injury (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Diffuse Alveolar Hemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
BK Virus Associated Hemorrhagic Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Adenovirus Viremia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
HSV Viremia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pseudomonas Aeruginosa Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Varicella Zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal GvHD (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Clostridium Difficile (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0
Pansinusitis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Renal Insufficiency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Enterococcus/ASTR Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory Syncytial Virus Upper Respiratory Illness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Aspergillus Terreus Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Alpha Hemolytic Strep Bacteremia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Epstein-Barr Virus Post-Transplant Lymphoproliferative Disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stem Cell Infusion (N=9) | Low Dose Donor T-Cells (N=3) | High Dose Donor T-Cells (N=4)
Allergic Reaction due to Campath (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Atrial Flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Undetermined etiology
Hypertension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Fluid Overload (Metabolism and nutrition disorders) | 6 (6) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 2 (3)
Mucositis (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 9 (9) | 3 (3) | 4 (4)
Tacrolimus Induced Renal Insufficiency (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0)
Elevated Alanine Aminotransferase (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 2 (2)
Elevated Bilirubin (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 1 (1)
Tacrolimus Induced Headaches (General disorders) | 2 (2) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fungal Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Campath Induced Hives (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin GvHD (Skin and subcutaneous tissue disorders) | 5 (6) | 2 (2) | 3 (4)
Campath Induced Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal GvHD (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Upper Gastrointestinal GvHD (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (4)
Liver GvHD (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (3)
Aspirated Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Elevated Alkaline Phosphatase (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Cytomegalovirus Antigenemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fungal Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Bleed (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus Reactivation (Infections and infestations) | 3 (3) | 3 (3) | 3 (3)
Viral Lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Enterococcus Faecalis Bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Adenovirus Viremia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ocular GvHD (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
HSV Oral Lesions (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenic Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Renal Insufficiency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Altered Mental Status Change (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Headaches (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Staphylococcus Epidermidis Bacteremia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridium Difficile Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Epstein-Barr Viremia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Multifocal Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes